CLINICAL TRIAL: NCT06419569
Title: Efficacy of High Power Laser Versus Low Level Laser in Ultrasonographic and Functional Outcomes in Patients With Knee Osteoarthritis
Acronym: OA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nabil Mahmoud Ismail Abdel-Aal, principle investigator nabil mahmoud ismail abdel-aal, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003450
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Knee Osteoarthritis
Keywords: High Power Laser; Low Level Laser; Ultrasonographic changes; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: high power laser and low level laser
Who Masked: Investigator, Outcomes Assessor
Masking Description: opaque sealed envelop
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- high power laser (Experimental): thirty patients will receive high-power laser and conventional physical therapy three times a week for eight weeks
  Interventions: Other: high power laser; Other: conventional physical therapy
- low level laser (Experimental): thirty patients will receive low level laser and conventional physical therapy three times a week for eight weeks
  Interventions: Other: low level laser; Other: conventional physical therapy
- conventional physical therapy (Active Comparator): thirty patients will receive conventional physical therapy three times a week for eight weeks
  Interventions: Other: conventional physical therapy

INTERVENTIONS:
Other: high power laser — Sessions will performed with scanning in longitudinal and perpendicular direction on the medial and lateral sides of the knee with Laser scanner machine. handpiece was positioned in contact and perpendicularly while the patient in a supine lying position with the knee flexed at 30° to open the joint surfaces to the laser beam (optical windows). The scanning was performed transversely and longitudinally in the anterior, medial, and lateral aspects of the knee joint with emphasis on the application on the joint line between the tibial and femoral epicondyles. The total energy delivered to the patient during one session was 1,250 J through three phases of treatment. The initial phase is performed with fast manual scanning with a total of 500 J. In the initial phase, the laser fluency is set to two successive subphases of 710 and 810 mJ/cm2 for a total of 500 J.
  Arms: high power laser
Other: low level laser — patients will receive laser with 0.5 W to gain energy density of 6 J/cm2, and total energy of 240 J during one session. LASER apparatus that will be used is Chattanoga Intelect Laser with 850nm wavelength and 200mW power Lasers. Same three phases like HPL with different energy dose. First phase: Fast manual scan 100 J. Second 10 point joint line phase with evey point 14 seconds and 4J to deliver a total of 40 J in this phase. Third phase: Slow manual scan 100 J.
  Arms: low level laser
Other: conventional physical therapy — the patients will receive conventiobal physical therapy in the form of Exercise therapy program (1) Warm-up exercises: Walking at the usual speed on a flat surface for 10 min with hamstring and calf gentle stretches.(2) Major exercises for knee OA: Straight leg raise, quadriceps setting, heel raise, one leg balance, step ups, and quadriceps strengthening exercises. The US protocol consists of continuous ultrasonic waves of 1 MHz frequency and 1 W/cm2 intensity applied with a 5-cm diameter applicator. The patients will be placed in a supine position, and the US applied to the medial and lateral parts (5 min on each side) of the knee in circular movements with the probe at right angles to ensure maximum absorption of the energy.

SUMMARY:
this study will be conducted to compare between high power laser and low-intensity laser on ultrasonographic and functional outcomes in patients with knee osteoarthritis

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a major source of pain, disability, and socioeconomic cost worldwide. The epidemiology of the disorder is complex and multifactorial, with genetic, biological, and biomechanical components. It is estimated that 63 to 85 percent of Americans over age 65 have radiographic signs of OA and that 35 to 50 percent have symptoms of pain, stiffness or limitation of motion. Between 9 and 12 percent of elderly Americans (approximately 3 million people) have enough impairment from OA that they cannot perform their major activities, and half of these individuals are totally disabled (confined to bed or a wheelchair). High power laser therapy (HPL) that involves higher-intensity laser radiation is a new, painless, and powerful modality that showed significant results in pain reduction. One of the modalities commonly used by clinicians was Low Level Laser Therapy introduced as an alternative, safe and non-invasive treatment for OA about 30 years ago.A more recent systemic review investigated the effects of low-level and high-intensity laser therapy as adjunctive to rehabilitation exercise on pain, stiffness and function in knee osteoarthritis and concluded that Both LLLT and HPL are beneficial as adjuncts to rehabilitation exercise in the management of knee OA. Based on an indirect comparison, the HPL and exercise seems to have higher efficacy in reducing knee pain and stiffness, and in increasing function. To confirm this finding, a direct comparative investigation of the two types of laser therapy may be necessary. ninety patients with knee osteoarthritis will be assigned randomly to three groups; the first experimental will receive high power laser plus conventional physical therapy, second one will receive low-intensity laser and traditional physical therapy, finally, the third group will receive traditionally therapy only

ELIGIBILITY:
Inclusion Criteria:

* X-ray stages II and III osteoarthritis
* Age between 45 and 75 years.
* BMI equal to or less than 35.

Exclusion Criteria:

* Unwillingness to participate in the study.
* Uncompleted evaluation/treatment programs.
* Any damage to the knee joint during the study.
* Using any treatment other than prescribed therapeutic protocols.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05-30 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
osteophyte diameter | up to eight weeks
  ultrasonographe device will be used to assess the osteophyte diameter
hyaline cartilage thickness assessment | up to eight weeks
  utrasonographe device will be used to assess hyaline cartilage thickness

SECONDARY OUTCOMES:
knee function | up to eight weeks
  Knee Injury and Osteoarthritis Outcome Score questionnaire will be used to assess knee function.five patient-relevant subscales of KOOS are scored separately: Pain (nine items); Symptoms (seven items); ADL Function (17 items); Sport and Recreation Function (five items); Quality of Life (four items). A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic assessment scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.
pain intensity | up to eight weeks
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. The following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm)
knee range of motion | up to eight weeks
  digital goniometer will be used to assess knee range of motion
pressure pain threshold | up to eight weeks
  algometer will be used to assess pressure pain threshold